CLINICAL TRIAL: NCT03488446
Title: Radiomics for Prediction of Lymph Node Metastasis in Gastric Cancer（RPLNM）(GIPMCS-1701)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); The Third Affiliated Hospital of Southern Medical University (Other Government)
Responsible Party: Sponsor
Other Study IDs: GIPMCS-1701
Record Dates: First submitted 2017-09-30; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2017-08

CONDITIONS: Digestive System Diseases; Gastrointestinal Neoplasms; Digestive System Neoplasms; Gastrointestinal Diseases; Stomach Neoplasms
Keywords: Gastric Cancer; Radiomics; Computed Tomograpy; Lymph Node Metastasis; Prediction
MeSH Terms: conditions — Digestive System Diseases; Gastrointestinal Neoplasms; Digestive System Neoplasms; Gastrointestinal Diseases; Stomach Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study proposes to establish a CT radiomics-based prediction model for identifying metastasis of each station lymph nodes in gastric cancer.

DETAILED DESCRIPTION:
This is a prospective, multi-center trial conducted at 4 high-volume gastric cancer centers in China (Nanfang Hospital of Southern Medical University; Sun Yat-Sen University Cancer Center; First Affiliated Hospital, Sun Yat-Sen University; The Third Affiliated Hospital, Sun Yat-Sen University) designed to determine the predicted performance of radiomics-based prediction model for identifying metastasis of each station lymph nodes by enhanced CT for preoperative noninvasive assessment of the lymph node status in patients with gastric cancer. The study includes the construction of CT radiomics-based prediction model and the validation of the prediction model.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years;
* Patients providing written informed consent;
* Pathologically proven gastric cancer scheduled to preoperative enhanced abdomen CT and undergo gastrectomy with type D2 lymphadenectomy;
* Has undergone > 64 multi-detector row CT within 14 days prior to surgical resection; .No receipt of preoperative therapy (radiotherapy, chemotherapy or chemoradiotherapy).

Exclusion Criteria:

* Preoperative therapy (radiotherapy, chemotherapy or chemoradiotherapy);
* Failed to receive preoperative enhanced abdomen CT or undergo gastrectomy with type D2 lymphadenectomy;
* Inavailable pathological results for local lymph node status;
* Inquality of CT images for feature extraction; .Patient quit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pathologically proven gastric cancer patients who receive preoperative CT and surgical resection in these hospitals.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-08-30 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Pathological lymph node status of every station | Pathologic evaluation will be performed for each patient within 1 week after surgery
  Pathological lymph node status of each station is defined as lymph node metastasis exist or not

SECONDARY OUTCOMES:
Survival time | Follow-up from the date of surgery to the date of death.
  Disease-free survival and overall survival
Lymph node stage (N stage) | Pathologic evaluation will be performed for each patient within 1 week after surgery
  Pathological lymph node stage after surgery (N0 stage: no lymph node metastassis; N1 stage: 1-2 lymph node metastasis; N2 stage: 3-6 lymph node metastasis; N3a stage: 7-15 lymph node metastasis;N3b stage: >15 lymph node metastassis)

CONTACTS AND LOCATIONS:
Overall Officials: Guoxin Li, M.D., PH.D., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Gillies RJ, Kinahan PE, Hricak H. Radiomics: Images Are More than Pictures, They Are Data. Radiology. 2016 Feb;278(2):563-77. doi: 10.1148/radiol.2015151169. Epub 2015 Nov 18. PMID 26579733
- [Result] Aerts HJ, Velazquez ER, Leijenaar RT, Parmar C, Grossmann P, Carvalho S, Bussink J, Monshouwer R, Haibe-Kains B, Rietveld D, Hoebers F, Rietbergen MM, Leemans CR, Dekker A, Quackenbush J, Gillies RJ, Lambin P. Decoding tumour phenotype by noninvasive imaging using a quantitative radiomics approach. Nat Commun. 2014 Jun 3;5:4006. doi: 10.1038/ncomms5006. PMID 24892406
- [Result] Huang YQ, Liang CH, He L, Tian J, Liang CS, Chen X, Ma ZL, Liu ZY. Development and Validation of a Radiomics Nomogram for Preoperative Prediction of Lymph Node Metastasis in Colorectal Cancer. J Clin Oncol. 2016 Jun 20;34(18):2157-64. doi: 10.1200/JCO.2015.65.9128. Epub 2016 May 2. PMID 27138577